CLINICAL TRIAL: NCT04244734
Title: Implementation of an Early Rehabilitation Program for the Patient With Lung Transplantation: From the ICU to Home.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR(AG)49-2019
Record Dates: First submitted 2020-01-17; First posted 2020-01-28 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Lung Transplant; Rehabilitation
Keywords: lung transplantation; rehabilitation; respiratory muscle training; early mobilisation; Neuromuscular electrostimulation; in-bed cycling

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): The control group receives regular treatment in the ICU, which includes muscle strengthening exercises, passive/assisted or active mobilizations, and respiratory physiotherapy with breathing muscle strengthening in a medium load (initially at 40% load from results in MIP).
  Interventions: Other: Usual care treatment
- Group 2 (Experimental): The experimental group receives a new early rehabilitation program based on a patient's in-bed cycling that allows controlled and adapted training to the patient's situation, along with coordinated exercise with neuromuscular electrostimulation and respiratory physiotherapy with breathing muscle strengthening in a high load (initially at 60% load from results in MIP).
  Interventions: Other: New Treatment Protocol-MotoMED®

INTERVENTIONS:
Other: Usual care treatment — All evaluations are the same in both groups:
  Baseline evaluation
  ICU admission (If patient hemodynamically stable initiates physiotherapy treatment within the first 15 days after surgery).
  Treatment:A daily session from Monday to Friday of 40 minutes according to patient functional status: Passive or active-assisted or active mobilizations, muscle enhancement, respiratory physiotherapy and inspiratory muscle training at 40% of the PIM value.
  2nd evaluation when patient has a RASS -1/0 score: 3rd evaluation when ICU discharge.
  Treatment ward: A 60-minute daily session according to patient functional status in the gym (physiotherapy area in hospital): Cycloergometer, muscle enhancement, respiratory physiotherapy and inspiratory muscle training.
  4th evaluation when hospital discharge 5th evaluation (1 month after discharge) 6th evaluation (4 months after discharge) 7th evaluation (1 year after surgery)
  Other Names: usual care
  Arms: Group 1
Other: New Treatment Protocol-MotoMED® — Baseline evaluation
  ICU admission (If patient hemodynamically stable initiates physiotherapy treatment within the first 15 days after surgery).
  Treatment: A daily session from Monday to Friday of 40 minutes (5 minutes of warm-up, 30 of training and 5 of cooling). Combined quadriceps / biceps femoris electrotherapy: at 200-350μs intensity. Respiratory physiotherapy with the objectives: Airway permeabilization and inspiratory muscle training at 60% of the PIM value.
  2nd evaluation when patient has a RASS -1/0 score: 3rd evaluation when ICU discharge.
  Treatment ward: A 60-minute daily session according to patient functional status in the gym (physiotherapy area in hospital): Cycloergometer, muscle enhancement, respiratory physiotherapy and inspiratory muscle training.
  4th evaluation when hospital discharge 5th evaluation (1 month after discharge) 6th evaluation (4 months after discharge) 7th evaluation (1 year after surgery)
  Other Names: MotoMED + NEMS
  Arms: Group 2

SUMMARY:
Introduction: Following pulmonary transplantation (PT), peripheral and respiratory muscle weakness, and associated global malfunction are some of the limiting factors in rapid recovery. Effective early implantation pulmonary rehabilitation programs are currently lacking.

Objectives: To introduce an early rehabilitation program in the ICU after PT to see if there is an improvement in functionality, an increase in strength and muscle mass, an improvement in the strength of the respiratory muscles and a shorter hospitalization time in the ICU and in the ward.

Methodology: A single-blind randomized clinical trial will be performed to divide patients with PT into one experimental group and another control group. Prior to the PT, those patients between the ages of 18 and 70 will be recruited, to be admitted to the ICU of Vall Hebron University Hospital, and who have been prescribed pulmonary rehabilitation with onset in the first 15 days after the surgery. The control group receives regular treatment in the ICU, which includes muscle strengthening exercises, passive/assisted or active mobilizations, and respiratory physiotherapy with breathing muscle strengthening in a medium load. The experimental group receives a new early rehabilitation program based on a patient's in-bed cycling that allows controlled and adapted training to the patient's situation, along with coordinated exercise with neuromuscular electrostimulation and respiratory physiotherapy with breathing muscle strengthening in a high load. Improvement will be observed through functional scales (6MWT), muscle dynamometry, manual muscle test (MRC-SumScore), bioimpedanciometry, inspiratory and maximal expiratory pressures, spirometry, frailty and sarcopenia tests and a long-term Cardiopulmonary Exercise Testing.

Expected Outcomes: Patients who perform the experimental group are expected to have an early discharge from the ICU and a reduction of the total hospital admission. Is also expected that the experimental group will improve the functional capacity and muscular strength, and they will have a lower risk of fragility in long term. It is also expected that the patients in the experimental group will soon be able to normalize their oxygen consumption a year after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral lung transplantation.
* Age criteria (From 18 to 70 years old).
* Start the rehabilitation program between the first 15 days after lung transplantation.

Exclusion Criteria:

* Do not meet inclusion criteria.
* Fulfill some criterion of absolute contraindication for the use of electrostimulation in the lower extremities (pacemaker, pregnancy or unstable fracture that requires absolute rest and immobilization.
* Cognitive or psychiatric alteration that does not allow you to participate in the project.
* Not wanting to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | Through study completion, an average of 1 year
  Measured with 6MWT
  It will be measured in different moments:
  Baseline Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge
Muscle strength | Through study completion, an average of 1 year
  Measured with dynamometer
  It will be measured in different moments
  Baseline When patient awake in ICU (RASS -1/0) Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge
Muscle mass | Through study completion, an average of 1 year
  Measured with bioimpedanciometry
  It will be measured in different moments:
  Baseline Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge
Respiratory muscle strength | Through study completion, an average of 1 year
  Measured with MIP and MEP
  It will be measured in different moments
  Baseline When patient awake in ICU (RASS -1/0) Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge
Cough strength | Through study completion, an average of 1 year
  Measured with Peak Cough Flow
  It will be measured in different moments
  Baseline When patient awake in ICU (RASS -1/0) Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge

SECONDARY OUTCOMES:
Frailty | Through study completion, an average of 1 year
  Measured with the short physical performance battery test (SPPB test)
  SPPB (maximum 12 points)
  * 7 points or less: Frailty
  * 8 to 9 points: Pre-frailty
  * More than 10 points: Not frailty
  It will be measured in different moments:
  Baseline Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge
Muscle balance | Through study completion, an average of 1 year
  Measured with the Medical Research Council sum score test
  It will be measured in different moments
  Baseline When patient awake in ICU (RASS -1/0) Hospital discharge After 1 month of discharge After 4 month of discharge
  1 year after the discharge
Pulmonary Capacity | Through study completion, an average of 1 year
  Measured with a spirometer
  We will interpret the data obtained from forced spirometry to evaluate how our patient's pulmonary functions is developing after the surgery.
  Data collection:
  FEV1/FVC: It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).The result of this ratio is expressed as FEV1%.
  The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
  It will be measured in different moments Baseline
  1 year after the discharge
Oxygen consumption | Through study completion, an average of 1 year
  Measured with the Cardiopulmonary effort test
  It will be measured in different moments
  After 1 month of discharge After 4 month of discharge
  1 year after the discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bernat Planas Pascual, PT, MSc, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute
Locations (1):
- Hospital Universitari Vall d'Hebron Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, King TE Jr, Lancaster L, Noble PW, Sahn SA, Thomeer M, Valeyre D, Wells AU. Forced vital capacity in patients with idiopathic pulmonary fibrosis: test properties and minimal clinically important difference. Am J Respir Crit Care Med. 2011 Dec 15;184(12):1382-9. doi: 10.1164/rccm.201105-0840OC. Epub 2011 Sep 22. PMID 21940789
- [Background] Roman A, Ussetti P, Sole A, Zurbano F, Borro JM, Vaquero JM, de Pablo A, Morales P, Blanco M, Bravo C, Cifrian J, de la Torre M, Gamez P, Laporta R, Monforte V, Mons R, Salvatierra A, Santos F, Sole J, Varela A; Sociedad Espanola de Neumologia y Cirugia Toracica. Guidelines for the selection of lung transplantation candidates. Arch Bronconeumol. 2011 Jun;47(6):303-9. doi: 10.1016/j.arbres.2011.03.007. Epub 2011 May 4. English, Spanish. PMID 21536362
- [Background] Coll E, Santos F, Ussetti P, Canela M, Borro JM, De La Torre M, Varela A, Zurbano F, Mons R, Morales P, Pastor J, Salvatierra A, de Pablo A, Gamez P, Moreno A, Sole J, Roman A. The Spanish Lung Transplant Registry: first report of results (2006-2010). Arch Bronconeumol. 2013 Feb;49(2):70-8. doi: 10.1016/j.arbres.2012.06.001. Epub 2012 Aug 28. English, Spanish. PMID 22939738
- [Background] Weill D, Benden C, Corris PA, Dark JH, Davis RD, Keshavjee S, Lederer DJ, Mulligan MJ, Patterson GA, Singer LG, Snell GI, Verleden GM, Zamora MR, Glanville AR. A consensus document for the selection of lung transplant candidates: 2014--an update from the Pulmonary Transplantation Council of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2015 Jan;34(1):1-15. doi: 10.1016/j.healun.2014.06.014. Epub 2014 Jun 26. PMID 25085497
- [Background] Weill D. Lung transplantation: indications and contraindications. J Thorac Dis. 2018 Jul;10(7):4574-4587. doi: 10.21037/jtd.2018.06.141. PMID 30174910
- [Background] Shigemura N, Bhama J, Gries CJ, Kawamura T, Crespo M, Johnson B, Zaldonis D, Pilewski J, Toyoda Y, Bermudez C. Lung transplantation in patients with prior cardiothoracic surgical procedures. Am J Transplant. 2012 May;12(5):1249-55. doi: 10.1111/j.1600-6143.2011.03946.x. Epub 2012 Feb 2. PMID 22300103
- [Background] Reynaud-Gaubert M, Mornex JF, Mal H, Treilhaud M, Dromer C, Quetant S, Leroy-Ladurie F, Guillemain R, Philit F, Dauriat G, Grenet D, Stern M. Lung transplantation for lymphangioleiomyomatosis: the French experience. Transplantation. 2008 Aug 27;86(4):515-20. doi: 10.1097/TP.0b013e31817c15df. PMID 18724219
- [Background] Detterbeck FC, Egan TM, Mill MR. Lung transplantation after previous thoracic surgical procedures. Ann Thorac Surg. 1995 Jul;60(1):139-43. PMID 7598576
- [Background] Curtis HJ, Bourke SJ, Dark JH, Corris PA. Lung transplantation outcome in cystic fibrosis patients with previous pneumothorax. J Heart Lung Transplant. 2005 Jul;24(7):865-9. doi: 10.1016/j.healun.2004.05.024. PMID 15982615
- [Background] American Thoracic Society. Idiopathic pulmonary fibrosis: diagnosis and treatment. International consensus statement. American Thoracic Society (ATS), and the European Respiratory Society (ERS). Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):646-64. doi: 10.1164/ajrccm.161.2.ats3-00. No abstract available. PMID 10673212
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, Lancaster L, Noble PW, Raghu G, Sahn SA, Szwarcberg J, Thomeer M, Valeyre D, King TE Jr. Ascertainment of individual risk of mortality for patients with idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 Aug 15;184(4):459-66. doi: 10.1164/rccm.201011-1790OC. PMID 21616999
- [Background] de Gracia J, Mata F, Alvarez A, Casals T, Gatner S, Vendrell M, de la Rosa D, Guarner L, Hermosilla E. Genotype-phenotype correlation for pulmonary function in cystic fibrosis. Thorax. 2005 Jul;60(7):558-63. doi: 10.1136/thx.2004.031153. PMID 15994263
- [Background] De Soyza A, Archer L, Wardle J, Parry G, Dark JH, Gould K, Corris PA. Pulmonary transplantation for cystic fibrosis: pre-transplant recipient characteristics in patients dying of peri-operative sepsis. J Heart Lung Transplant. 2003 Jul;22(7):764-9. doi: 10.1016/s1053-2498(02)00641-1. PMID 12873544
- [Background] Rosenbluth DB, Wilson K, Ferkol T, Schuster DP. Lung function decline in cystic fibrosis patients and timing for lung transplantation referral. Chest. 2004 Aug;126(2):412-9. doi: 10.1378/chest.126.2.412. PMID 15302726
- [Background] A.R.Damasio. The New England Journal of Medicine Downloaded from nejm.org at the Bodleian Libraries of the University of Oxford on February 16, 2014. For personal use only. No other uses without permission. Copyright © 1992 Massachusetts Medical Society. All rights re. N Engl J Med. 1992;327(26):1832-5.
- [Background] Mayer-Hamblett N, Rosenfeld M, Emerson J, Goss CH, Aitken ML. Developing cystic fibrosis lung transplant referral criteria using predictors of 2-year mortality. Am J Respir Crit Care Med. 2002 Dec 15;166(12 Pt 1):1550-5. doi: 10.1164/rccm.200202-087OC. Epub 2002 Aug 15. PMID 12406843
- [Background] Liou TG, Adler FR, Huang D. Use of lung transplantation survival models to refine patient selection in cystic fibrosis. Am J Respir Crit Care Med. 2005 May 1;171(9):1053-9. doi: 10.1164/rccm.200407-900OC. Epub 2005 Feb 1. PMID 15695493
- [Background] Ellaffi M, Vinsonneau C, Coste J, Hubert D, Burgel PR, Dhainaut JF, Dusser D. One-year outcome after severe pulmonary exacerbation in adults with cystic fibrosis. Am J Respir Crit Care Med. 2005 Jan 15;171(2):158-64. doi: 10.1164/rccm.200405-667OC. Epub 2004 Oct 22. PMID 15502116
- [Background] Kim D, George MP. Pulmonary Hypertension. Med Clin North Am. 2019 May;103(3):413-423. doi: 10.1016/j.mcna.2018.12.002. PMID 30955510
- [Background] Hoeper MM, Bogaard HJ, Condliffe R, Frantz R, Khanna D, Kurzyna M, Langleben D, Manes A, Satoh T, Torres F, Wilkins MR, Badesch DB. Definitions and diagnosis of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D42-50. doi: 10.1016/j.jacc.2013.10.032. PMID 24355641
- [Background] Handoko ML, Lamberts RR, Redout EM, de Man FS, Boer C, Simonides WS, Paulus WJ, Westerhof N, Allaart CP, Vonk-Noordegraaf A. Right ventricular pacing improves right heart function in experimental pulmonary arterial hypertension: a study in the isolated heart. Am J Physiol Heart Circ Physiol. 2009 Nov;297(5):H1752-9. doi: 10.1152/ajpheart.00555.2009. Epub 2009 Sep 4. PMID 19734361